CLINICAL TRIAL: NCT00645619
Title: Use of a Novel Protein (sTREM-1) to Differentiate Pure Viral Lung Infection From Viral With Co-existing Bacterial Lung Infection
Brief Title: Use of TREM-1 Protein to Differentiate Viral and Bacterial Pneumonias in Intubated Children
Status: Withdrawn | Type: Observational
Why Stopped: PI is no longer with the University
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 022007-022
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Viral Pneumonia; Bacterial Pneumonia
Keywords: Pneumonia,viral; Pneumonia,bacterial; TREM-1 protein,human
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage fluid and Serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients with pure viral pneumonia
- 2: Patients with viral pneumonia along with secondary bacterial pneumonia
- 3: Patients with significant bacterial pneumonia
- 4: Patients with congenital heart disease undergoing cardiopulmonary bypass who have no pneumonia

SUMMARY:
The purpose of this study is to determine whether a protein called TREM-1 can be used to differentiate viral and bacterial pneumonias in children who are on ventilator support. We propose that the level of TREM-1 will be significantly elevated in the lung fluid of children with bacterial pneumonia and viral with co-existing bacterial pneumonia than in children with pure viral pneumonia.

DETAILED DESCRIPTION:
Most often, viruses are the cause of pneumonia in children. However, viral pneumonias are frequently associated with secondary bacterial pneumonia. It is important, though difficult, to differentiate patients who only have viral pneumonia from those who have viral pneumonia with secondary bacterial pneumonia. This will help physicians to prescribe antibiotics to only those with bacterial pneumonia and avoid antibiotic use in those with pure viral pneumonia, thus help to limit health-care cost and to decrease emergence of antibiotic resistance. In adult studies, TREM-1 has been shown to be specifically expressed in bacterial infections.

We propose that measuring TREM-1 in the bronchoalveolar lavage (BAL) fluid will help to differentiate these groups. Our hypothesis is that concentration of TREM-1 will be significantly elevated in the BAL fluid of children with bacterial pneumonia and viral with co-existing bacterial pneumonia than in children with pure viral pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Children from birth to 18 years intubated for respiratory failure or for surgery as mentioned above within 48 hours of intubation.

Exclusion Criteria:

* Use of antibiotics >72 hours preceding the study (not applicable to the definite bacterial pneumonia group)
* Use of oral/parenteral glucocorticoid therapy <2 weeks prior to admission
* Presence of tracheostomy
* Active treatment for pulmonary arterial hypertension
* Mechanical ventilation with FIO2 >0.6, MAP>20
* Presence of severe pulmonary interstitial emphysema, pneumothorax, bradycardia (heart rate, <80 beats/min in neonates, <70 beats/min in infants), hypotension (mean arterial pressure, <40 mm Hg in neonates, <50 mm Hg in infants), and platelet count of <30,000/mm3.
* Immunodeficient or immunocompromised due to other conditions.
* Enrollment in another interventional study that employs BAL.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Intubated patients in the intensive care unit with respiratory failure. Intubated patients patients in the OR undergoing video-assisted thoracic surgery for empyema.
  Intubated patients undergoing cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03-24 (Estimated); Primary Completion 2008-03-26 (Estimated); Study Completion 2008-03-26 (Actual)

PRIMARY OUTCOMES:
TREM-1 level in the BAL fluid of patients with pure viral pneumonia in comparison to patients with viral with co-existing bacterial pneumonia | Within 48 hours of being intubated

SECONDARY OUTCOMES:
TREM-1 level in the BAL fluid of patients with pure bacterial pneumonia and no pneumonia | Within 48 hours of intubation for TREM-1 level
TREM-1 level in the serum of all 4 groups | Within 48 hours of intubation for TREM-1 level
Length of ventilator support, length of ICU and hospital stay | Within 48 hours of intubation for TREM-1 level

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hardy, MD, Study Director — University of Texas Southwestern Medical Center; Peter Luckett, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Childrens Medical Center, Dallas, Texas, United States